CLINICAL TRIAL: NCT04689906
Title: In-hospital Delay of Surgery Increases the Rate of Complicated Appendicitis in Patients Presenting With Short Duration of Symptoms: a Retrospective Cohort Study
Brief Title: Patient Time and In-hospital Delay of Surgery Association With Complicated Appendicitis
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Itamar Ashkenazi MD, Staff Physician, Rambam Health Care Campus
Other Study IDs: HTVSPTAPP1
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Acute Appendicitis
Keywords: Appendicitis; Ruptured Appendicitis; Appendectomy; Timing of Surgery
MeSH Terms: conditions — Appendicitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: surgery — This is a retrospective study that includes patients operated for suspicion of acute appendicitis

SUMMARY:
This is a retrospective observational study with its main aim of evaluating possible factors associated with complicated appendicitis. Current literature supports time from symptom onset until registration as the main and maybe only determinant of the outcome if patients are operated on within 24 hours. We wish to evaluate whether this is true in all patients, or there are subgroups in which time from registration to operation is associated with complicated appendicitis.

DETAILED DESCRIPTION:
The data to be analyzed is that of patients operated on acutely for suspected appendicitis within 10 years in one medical center. Patients undergoing interval or incidental appendectomies will not be included. The endpoint to be evaluated is complicated appendicitis (gangrenous, abscess, perforated). The independent variables will include mainly sex, age, patient time (time from symptom onset to registration), hospital time (time from registration to operation), and missed diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients of all ages who underwent appendectomy of acute appendicitis in a single medical center between December 1, 2006, and December 31, 2016

Exclusion Criteria:

* interval appendectomy,
* incidental appendectomy,
* appendectomy after failed antibiotic treatment for either acute appendicitis or peri-appendicular abscess
* patients with a non-inflamed appendix
* those in whom symptom onset before hospitalization was not noted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated in one medical center during one decade.
Sampling Method: Non-Probability Sample
Enrollment: 3137 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
proportion of complicated appendicitis | finding during surgery/pathology
  complicated appendicitis defined as either gangrenous appendicitis, perforation with abscess, perforation with local peritonitis, perforation with diffuse peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Ashkenazi, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available upon reasonable request

REFERENCES:
- [Background] Ashkenazi I, Zeina AR, Olsha O. Early ultrasound in acute appendicitis avoids CT in most patients but delays surgery and increases complicated appendicitis if nondiagnostic - A retrospective study. Am J Surg. 2020 Apr;219(4):683-689. doi: 10.1016/j.amjsurg.2019.05.013. Epub 2019 May 25. PMID 31153584
- [Derived] Ashkenazi I, Zeina AR, Olsha O. In-hospital delay of surgery increases the rate of complicated appendicitis in patients presenting with short duration of symptoms: a retrospective cohort study. Eur J Trauma Emerg Surg. 2022 Oct;48(5):3879-3886. doi: 10.1007/s00068-022-01912-3. Epub 2022 Feb 24. PMID 35211772